CLINICAL TRIAL: NCT03355742
Title: XIENCE 28 Global Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10235
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Bleeding Disorder; Stroke, Ischemic; Stroke Hemorrhagic; Hematological Disease; Thrombocytopenia; Coagulation Disorder; Anemia; Renal Insufficiency; Coronary Artery Disease
Keywords: XIENCE; High bleeding risk (HBR); Dual antiplatelet therapy (DAPT); Coronary Artery Disease; Drug eluting stent (DES)
MeSH Terms: conditions — Hemostatic Disorders; Ischemic Stroke; Hemorrhagic Stroke; Hematologic Diseases; Thrombocytopenia; Anemia; Renal Insufficiency; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- XIENCE (Experimental): XIENCE + Short duration (1 month) of DAPT
  Interventions: Device: XIENCE; Drug: DAPT

INTERVENTIONS:
Device: XIENCE — Subjects who received XIENCE family stent systems will be included.
Drug: DAPT — 1-month clear subjects will receive 1 month of P2Y12 inhibitor and 12 months of aspirin after index procedure.
  Other Names: Dual antiplatelet therapy

SUMMARY:
XIENCE 28 Global Study is a prospective, single arm, multi-center, open label, non-randomized trial to further evaluate the safety of 1-month (as short as 28 days) dual antiplatelet therapy (DAPT) in subjects at high risk of bleeding (HBR) undergoing percutaneous coronary intervention (PCI) with the approved XIENCE family (XIENCE Xpedition Everolimus Eluting Coronary Stent System [EECSS], XIENCE Alpine EECSS, XIENCE PROX EECSS, XIENCE ProA EECSS or XIENCE Sierra EECSS of coronary drug-eluting stents

DETAILED DESCRIPTION:
The XIENCE 28 Global Study will evaluate the safety of 1-month DAPT following XIENCE implantation in HBR patients. A minimum of 800 to a maximum of 960 subjects will be registered from approximately 50 sites globally and subject registration is capped at 120 per site. Eligibility of P2Y12 receptor inhibitor discontinuation will be assessed at 1-month follow-up. Subjects who are free from myocardial infarction (MI), repeat coronary revascularization, stroke, or stent thrombosis (ARC definite/probable) within 1 month (prior to 1-month visit but at least 28 days) after stenting and have been compliant with 1-month DAPT without interruption of either aspirin and/or P2Y12 receptor inhibitor for > 7 consecutive days are considered as "1-month clear", and will discontinue P2Y12 receptor inhibitor as early as 28 days and continue with aspirin monotherapy through 12-month follow-up.

All registered subjects will be followed at 1, 3, 6 and 12 months post index procedure. The data collected from the XIENCE 28 Global Study will be compared with the historical control of non-complex HBR subjects treated with standard DAPT up to 12 months from the XIENCE V USA Study .

ELIGIBILITY:
Inclusion Criteria:

1. Subject is considered at HBR, defined as meeting one or more of the following criteria at the time of registration and in the opinion of the referring physician, the risk of major bleeding with > 1-month DAPT outweighs the benefit:

   1. Subjects ≥ 75 years of age.
   2. Clinical indication for chronic (at least 6 months) or lifelong anticoagulation therapy.
   3. History of major bleeding which required medical attention within 12 months of the index procedure.
   4. History of stroke (ischemic or hemorrhagic).
   5. Renal insufficiency (creatinine ≥ 2.0 mg/dl) or failure (dialysis dependent).
   6. Systemic conditions associated with an increased bleeding risk (e.g. hematological disorders, including a history of or current thrombocytopenia defined as a platelet count <100,000/mm^3, or any known coagulation disorder associated with increased bleeding risk).
   7. Anemia with hemoglobin < 11g/dl.
2. Subject must be at least 18 years of age.
3. Subject must provide written informed consent as approved by the Ethics Committee (EC) of the respective clinical site prior to any trial related procedure.
4. Subject is willing to comply with all protocol requirements, including agreement to stop taking P2Y12 inhibitor at 1 month, if eligible per protocol.
5. Subject must agree not to participate in any other clinical trial for a period of one year following the index procedure.

Angiographic Inclusion Criteria

1. Up to three target lesions with a maximum of two target lesions per epicardial vessel.

   Note:
   1. The definition of epicardial vessels means left anterior descending coronary artery (LAD), left circumflex coronary artery (LCX) and right coronary artery (RCA) and their branches. For example, the subject must not have >2 lesions requiring treatment within both the LAD and a diagonal branch in total.
   2. If there are two target lesions within the same epicardial vessel, the two target lesions must be at least 15 mm apart per visual estimation; otherwise this is considered as a single target lesion.
2. Target lesion must be located in a native coronary artery with visually estimated reference vessel diameter between 2.25 mm and 4.25 mm.
3. Exclusive use of XIENCE family of stent systems during the index procedure.
4. Target lesion has been treated successfully, which is defined as achievement of a final in-stent residual diameter stenosis of <20% with final thrombolysis in myocardial infarction (TIMI-3) flow assessed by online quantitative angiography or visual estimation, with no residual dissection National Heart, Lung, and Blood Institute (NHLBI) grade ≥ type B, and no transient or sustained angiographic complications (e.g., distal embolization, side branch closure), no chest pain lasting > 5 minutes, and no ST segment elevation > 0.5mm or depression lasting > 5 minutes.

Exclusion Criteria:

1. Subject with an indication for the index procedure of acute ST-segment elevation MI (STEMI).
2. Subject has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, P2Y12 inhibitors (clopidogrel/prasugrel/ticagrelor), everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
3. Subject with implantation of another drug-eluting stent (other than XIENCE) within 12 months prior to index procedure.
4. Subject has a known left ventricular ejection fraction (LVEF) <30%.
5. Subject judged by physician as inappropriate for discontinuation from P2Y12 inhibitor use at 1 month, due to another condition requiring chronic P2Y12 inhibitor use.
6. Subject with planned surgery or procedure necessitating discontinuation of P2Y12 inhibitor within 1 month following index procedure.
7. Subject with a current medical condition with a life expectancy of less than 12 months.
8. Subject intends to participate in an investigational drug or device trial within 12 months following the index procedure.
9. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.

   Note: Female subjects of childbearing potential should be instructed to use safe contraception (e.g., intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches hormonal vaginal devices, injections with prolonged release). It is accepted, in certain cases, to include subjects having a sterilised regular partner or subjects using a double barrier contraceptive method. However, this should be explicitly justified in special circumstances arising from the trial design, product characteristics and/or trial population.
10. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
11. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.

Angiographic Exclusion Criteria

1. Target lesion is in a left main location.
2. Target lesion is located within an arterial or saphenous vein graft.
3. Target lesion is restenotic from a previous stent implantation.
4. Target lesion is a chronic total occlusion (CTO, defined as lesion with TIMI flow 0 for at least 3 months).
5. Target lesion is implanted with overlapping stents, whether planned or for bailout.

Note: If there is more than one target lesion, all target lesions must satisfy the angiographic eligibility criteria. Non-target lesion (i.e., lesions that do not meet the angiographic criteria listed above) treatments are not allowed during the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 963 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, MD, Principal Investigator — Bern University Hospital
Locations (52):
- Kepler Universitätsklinikum GmbH, Linz, UPR AUS, Austria
- Belgium (4):
  - Onze-Lieve-Vrouwziekenhuis Campus Aalst, Aalst, Eflndrs
  - UZ Gent, Ghent, Flemish
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Jesse Ziekenhuis, Hasselt, Limburg
- China (2):
  - Beijing AnZhen Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Jilin University, Changchun, N China
- Germany (7):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen, Bad-wur
  - Elisabeth-Krankenhaus Essen GmbH, Essen, N. RHIN
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz, Rhinela
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Segeberger Kliniken GmbH, Bad Segeberg, Schlesw
  - Universitätsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - UKE Hamburg (Universitatsklinik Eppendorf), Hamburg
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong, Hong Ko
  - Queen Elizabeth Hospital, Hong Kong, Hong Ko
  - The University of Hong Kong (Queen Mary Hospital), Hong Kong, HONG KO
- Italy (8):
  - Clinica Mediterranea, Napoli, Campani
  - AOU Federico II - Università degli Studi di Napoli, Napoli, Campani
  - Az.Osp. Universitaria di Ferrara, Cona, Emi-rom
  - AOU di Parma, Parma, Emi-rom
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Rome, Lazio
  - Policlinico Universitario A. Gemelli, Rome, Lazio
  - Centro Cardiologico Monzino, Milan, Lombard
  - Istituto Clinico Humanitas, Rozzano, Lombard
- Netherlands (3):
  - Scheperziekenhuis, Emmen, Drenthe
  - Medisch Centrum Leeuwarden, Leeuwarden, Friesld
  - Albert Schweitzer Ziekenhuis, Dordrecht, ZUID
- Portugal (2):
  - Hospital de Santa Cruz, Carnaxide, Lisbon District
  - Santa Maria Hospital, Lisbon, Lisbon District
- Singapore (2):
  - National Heart Centre Singapore, Singapore, Central
  - Tan Tock Seng Hospital, Singapore, Central
- Spain (7):
  - HCU Virgen de la Victoria, Málaga, Andalu
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabr
  - Hospital del Mar, Barcelona, Catalon
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Catalon
  - Hospital Clinico Universitario de Valladolid, Valladolid, Cstleon
  - Hospital Alvaro Cunqueiro Dept of Interventional Cardiology, Vigo, Pontev
  - Hospital Universitario Doce de Octubre, Madrid
- Switzerland (3):
  - Kantonsspital Aarau, Aarau, Basel
  - Center Inselspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne
- Taiwan (4):
  - Chang Gung Memorial Hospital, Linkou District, Ntaiwan
  - National Taiwan University Hospital, Taipei, Ntaiwan
  - Taipei Veterans General Hospital (VGH), Taipei, Ntaiwan
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Staiwan
- United Kingdom (6):
  - Freeman Hospital, Newcastle upon Tyne, NE ENGL
  - Craigavon Area Hospital, Portadown, Nirelnd
  - Southampton University Hospital, Southampton, Soeast
  - Royal Bournemouth Hospital, Bournemouth, Sowest
  - Royal Devon and Exeter Hospital, Exeter, Sowest
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Derived] Valgimigli M, Cao D, Angiolillo DJ, Bangalore S, Bhatt DL, Ge J, Hermiller J, Makkar RR, Neumann FJ, Saito S, Picon H, Toelg R, Maksoud A, Chehab BM, Choi JW, Campo G, De la Torre Hernandez JM, Kunadian V, Sardella G, Thiele H, Varenne O, Vranckx P, Windecker S, Zhou Y, Krucoff MW, Ruster K, Zheng Y, Mehran R; XIENCE 90 and XIENCE 28 Investigators. Duration of Dual Antiplatelet Therapy for Patients at High Bleeding Risk Undergoing PCI. J Am Coll Cardiol. 2021 Nov 23;78(21):2060-2072. doi: 10.1016/j.jacc.2021.08.074. PMID 34794687
- [Derived] Valgimigli M, Cao D, Makkar RR, Bangalore S, Bhatt DL, Angiolillo DJ, Saito S, Ge J, Neumann FJ, Hermiller J, Picon H, Toelg R, Maksoud A, Chehab BM, Wang LJ, Wang J, Mehran R. Design and rationale of the XIENCE short DAPT clinical program: An assessment of the safety of 3-month and 1-month DAPT in patients at high bleeding risk undergoing PCI with an everolimus-eluting stent. Am Heart J. 2021 Jan;231:147-156. doi: 10.1016/j.ahj.2020.09.019. Epub 2020 Oct 6. PMID 33031789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 963 subjects were enrolled across 52 sites globally, between 09 February, 2018 and 30 April, 2020. The last subject last visit was on 30 April, 2020 and the final data was extracted from the database on 01 July, 2020.
Period: Overall Study
Arm/Group | XIENCE
Started | 963
Completed | 864
Not Completed | 99
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 29
Not completed — Physician Decision | 6
Not completed — Death | 55
Not completed — Administrative Closure of the Study, Other Status Change Reason, Missed Visit, Protocol Violation | 5

BASELINE CHARACTERISTICS:
Arm/Group | XIENCE
Number analyzed (Participants) | 963
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.84 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 320
  Male | 643
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 145
  Not Hispanic or Latino | 360
  Unknown or Not Reported | 458
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 124
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 381
  More than one race | 0
  Unknown or Not Reported | 458
Region of Enrollment [Number; unit: participants]
  Singapore | 22
  Hong Kong | 48
  United Kingdom | 30
  Portugal | 8
  Switzerland | 37
  Spain | 89
  Austria | 3
  Netherlands | 49
  Belgium | 64
  China | 7
  Taiwan | 48
  Italy | 231
  Germany | 327
Prior Percutaneous Coronary Intervention (PCI) [Number; unit: participants] | 276
History of Major Bleeding [Number; unit: participants] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  participants
    number analyzed (Participants) | 961
    (all) | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of Net Adverse Clinical Endpoint (NACE), by Propensity Score Quintiles
Description: Net Adverse Clinical Endpoint (NACE):
  A composite rate of all-cause death, all myocardial infarction (modified Academic Research Consortium [ARC]), stent thrombosis (ARC definite or probable), stroke or major bleeding (Bleeding defined by the Bleeding Academic Research Consortium [BARC] type 2-5)
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who completed follow up at the given time point. Subjects who were lost to follow-up or withdrew consent prior to that time point, without the endpoint of interest, are excluded from the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants
  Q1: number analyzed (Participants) | 15
  Q1 | 2
  Q2: number analyzed (Participants) | 55
  Q2 | 5
  Q3: number analyzed (Participants) | 124
  Q3 | 10
  Q4: number analyzed (Participants) | 245
  Q4 | 15
  Q5: number analyzed (Participants) | 389
  Q5 | 40

2. Secondary Outcome: Number of Participants With Composite of Net Adverse Clinical Endpoint (NACE)
Description: as for outcome 1
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 55

3. Secondary Outcome: Number of Participants With Composite of Net Adverse Clinical Endpoint (NACE)
Description: as for outcome 1
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 121

4. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definite/Probable, ARC Definite)
Description: Definite stent thrombosis:
  Definite stent thrombosis is considered to have occurred by either angiographic or pathologic confirmation.
  Probable stent thrombosis:
  Clinical definition of probable stent thrombosis is considered to have occurred after intracoronary stenting in the following cases:
  * Any unexplained death within the first 30 days
  * Irrespective of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who completed follow up at the given time point. Subjects who were lost to follow-up, or withdrew consent, or died before time point analyzed, without any Stent Thrombosis event, are excluded from the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 816
Participants | 4

5. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definite/Probable, ARC Definite)
Description: as for outcome 4
Time Frame: From 6 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 791
Participants | 0

6. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definite/Probable, ARC Definite)
Description: as for outcome 4
Time Frame: From 1 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 793
Participants | 4

7. Secondary Outcome: Number of Participants With All Death, Cardiac Death, Vascular Death, Non-cardiovascular Death
Description: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants | 13

8. Secondary Outcome: Number of Participants With All Death, Cardiac Death, Vascular Death, Non-cardiovascular Death
Description: as for outcome 7
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 30

9. Secondary Outcome: Number of Participants With All Death, Cardiac Death, Vascular Death, Non-cardiovascular Death
Description: as for outcome 7
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 43

10. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI) and MI Attributed to Target Vessel (TV-MI, Modified ARC)
Description: Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality)
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI:
    * Within 48h after PCI: CK-MB >3 x URL or Troponin > 3 x URL with baseline value < URL
    * Within 72h after CABG: CK-MB >5 x URL or Troponin > 5 x URL with baseline value < URL
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants | 16

11. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI) and MI Attributed to Target Vessel (TV-MI, Modified ARC)
Description: as for outcome 10
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 11

12. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI) and MI Attributed to Target Vessel (TV-MI, Modified ARC)
Description: as for outcome 10
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 27

13. Secondary Outcome: Number of Participants With Composite of Cardiac Death or MI (Modified ARC)
Description: Cardiac death:
  Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  MI (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality)
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI:
    * Within 48h after PCI: CK-MB >3 x URL or Troponin > 3 x URL with baseline value < URL
    * Within 72h after CABG: CK-MB >5 x URL or Troponin > 5 x URL with baseline value < URL
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants | 22

14. Secondary Outcome: Number of Participants With Composite of Cardiac Death or MI (Modified ARC)
Description: as for outcome 13
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 23

15. Secondary Outcome: Number of Participants With Composite of Cardiac Death or MI (Modified ARC)
Description: as for outcome 13
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 45

16. Secondary Outcome: Number of Participants With Composite of All Death or All MI (Modified ARC)
Description: All death: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  MI (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality)
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants | 29

17. Secondary Outcome: Number of Participants With Composite of All Death or All MI (Modified ARC)
Description: as for outcome 16
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 41

18. Secondary Outcome: Number of Participants With Composite of All Death or All MI (Modified ARC)
Description: as for outcome 16
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 70

19. Secondary Outcome: Number of Participants With All Stroke, Ischemic Stroke and Hemorrhagic Stroke
Description: An acute symptomatic episode of neurological dysfunction attributed to a vascular cause lasting more than 24 hours or lasting 24 hours or less with a brain imaging study or autopsy showing new infarction.
  * Ischemic Stroke: An acute symptomatic episode of focal cerebral, spinal, or retinal dysfunction caused by an infarction of central nervous system tissue.
  * Hemorrhagic Stroke: An acute symptomatic episode of focal or global cerebral or spinal dysfunction caused by a non-traumatic intraparenchymal, intraventricular, or subarachnoid hemorrhage.
  * Undetermined Stroke: A stroke with insufficient information to allow categorization as ischemic or hemorrhagic.
  * Pharmacologic, i.e., thrombolytic drug administration, or Non-pharmacologic, i.e., neurointerventional procedure (e.g., intracranial angioplasty)
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 815
Participants | 3

20. Secondary Outcome: Number of Participants With All Stroke, Ischemic Stroke and Hemorrhagic Stroke
Description: as for outcome 19
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 784
Participants | 3

21. Secondary Outcome: Number of Participants With All Stroke, Ischemic Stroke and Hemorrhagic Stroke
Description: as for outcome 19
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 785
Participants | 6

22. Secondary Outcome: Number of Participants With Clinically-indicated Target Lesion Revascularization (CI-TLR)
Description: TLR is defined as any repeat percutaneous intervention of the target lesion (the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent) or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as clinically indicated [CI] or not CI by the investigator prior to repeat angiography.
  A revascularization is considered CI if angiography at follow-up shows a percent diameter stenosis ≥ 50% and if any one below occurs:
  * A positive history of recurrent angina pectoris, presumably related to the target vessel;
  * Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  * Abnormal results of any invasive functional diagnostic test (e.g: Doppler flow velocity reserve, fractional flow reserve);
  * A TLR with a diameter stenosis ≥70% in the absence of the above mentioned ischemic signs or symptoms.
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants | 7

23. Secondary Outcome: Number of Participants With Clinically-indicated Target Lesion Revascularization (CI-TLR)
Description: as for outcome 22
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 3

24. Secondary Outcome: Number of Participants With Clinically-indicated Target Lesion Revascularization (CI-TLR)
Description: as for outcome 22
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 10

25. Secondary Outcome: Number of Participants With Clinically-indicated Target Vessel Revascularization (CI-TVR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself
  A revascularization is considered clinically indicated if angiography at follow-up shows a percent diameter stenosis ≥ 50% and if one of the following occurs:
  * A positive history of recurrent angina pectoris, presumably related to the target vessel;
  * Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  * Abnormal results of any invasive functional diagnostic test (e.g., Doppler flow velocity reserve, fractional flow reserve);
  * A TVR with a diameter stenosis ≥70% in the absence of the above mentioned ischemic signs or symptoms.
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants | 5

26. Secondary Outcome: Number of Participants With Clinically-indicated Target Vessel Revascularization (CI-TVR)
Description: as for outcome 25
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 4

27. Secondary Outcome: Number of Participants With Clinically-indicated Target Vessel Revascularization (CI-TVR)
Description: as for outcome 25
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 9

28. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF, Composite of Cardiac Death, TV-MI and CI-TLR)
Description: TLF is defined as a composite of all cardiac death, myocardial infarction attributed to target vessel or clinically-indicated TLR.
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants | 21

29. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF, Composite of Cardiac Death, TV-MI and CI-TLR)
Description: as for outcome 28
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 21

30. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF, Composite of Cardiac Death, TV-MI and CI-TLR)
Description: as for outcome 28
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 42

31. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF, a Composite of Cardiac Death, TV-MI and CI-TVR)
Description: TVF is defined as a composite of cardiac death, MI attributed to target vessel, clinically-indicated TLR, or clinically-indicated TVR, non-TLR.
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 828
Participants | 22

32. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF, a Composite of Cardiac Death, TV-MI and CI-TVR)
Description: as for outcome 31
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 811
Participants | 22

33. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF, a Composite of Cardiac Death, TV-MI and CI-TVR)
Description: as for outcome 31
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 825
Participants | 44

34. Secondary Outcome: Number of Participants With Bleeding Defined by the Bleeding Academic Research Consortium (BARC) Type 2-5 and Type 3-5
Description: Bleeding per Bleeding Academic Research Consortium (BARC)definitions are as follows:
  Type 0
  Type 1
  Type 2
  Type 3
  Type 4
  Type 5
  Where, Type 0 indicates no bleeding and type 5 indicates fatal bleeding.
Time Frame: From 1 to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 817
Participants
  BARC Type 2-5 | 44
  BARC Type 3-5 | 20

35. Secondary Outcome: Number of Participants With Bleeding Defined by the BARC, Type 2-5 and Type 3-5
Description: as for outcome 34
Time Frame: From 6 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 789
Participants
  BARC Type 2-5 | 19
  BARC Type 3-5 | 7

36. Secondary Outcome: Number of Participants With Bleeding Defined by BARC, Type 2-5 and Type 3-5
Description: as for outcome 34
Time Frame: From 1 to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 792
Participants
  BARC Type 2-5 | 61
  BARC Type 3-5 | 27

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | XIENCE
All-Cause Mortality (participants affected / at risk) | 55/963
Serious Adverse Events (participants affected / at risk) | 374/963
Other Adverse Events (participants affected / at risk) | 357/963
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE (N=963)
Anaemia (Blood and lymphatic system disorders) | 11
Bicytopenia (Blood and lymphatic system disorders) | 1
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 1
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1
Angina Pectoris (Cardiac disorders) | 55
Angina Unstable (Cardiac disorders) | 1
Aortic Valve Incompetence (Cardiac disorders) | 2
Aortic Valve Stenosis (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 27
Atrial Flutter (Cardiac disorders) | 3
Atrial Tachycardia (Cardiac disorders) | 1
Atrioventricular Block (Cardiac disorders) | 2
Atrioventricular Block Complete (Cardiac disorders) | 3
Atrioventricular Block Second Degree (Cardiac disorders) | 1
Bifascicular Block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 3
Cardiac Failure (Cardiac disorders) | 30
Cardiac Failure Acute (Cardiac disorders) | 6
Cardiac Failure Congestive (Cardiac disorders) | 4
Cardiac Tamponade (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Congestive Cardiomyopathy (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 7
Dressler's Syndrome (Cardiac disorders) | 1
Mitral Valve Incompetence (Cardiac disorders) | 5
Myocardial Infarction (Cardiac disorders) | 18
Myocardial Ischaemia (Cardiac disorders) | 1
Myopericarditis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pleuropericarditis (Cardiac disorders) | 1
Right Ventricular Failure (Cardiac disorders) | 1
Sick Sinus Syndrome (Cardiac disorders) | 3
Sinoatrial Block (Cardiac disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 2
Supraventricular Tachycardia (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 4
Tricuspid Valve Incompetence (Cardiac disorders) | 2
Ventricular Extrasystoles (Cardiac disorders) | 3
Ventricular Fibrillation (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 5
Vertigo (Ear and labyrinth disorders) | 3
Vertigo Positional (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Retinal Artery Occlusion (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Colonic Polyp (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 2
Faeces Discoloured (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis Erosive (Gastrointestinal disorders) | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Inguinal Hernia (Gastrointestinal disorders) | 2
Intestinal Ischaemia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 5
Death (General disorders) | 15
General Physical Health Deterioration (General disorders) | 1
Hernia Obstructive (General disorders) | 1
Impaired Healing (General disorders) | 1
Multi-Organ Failure (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 3
Cholangitis (Hepatobiliary disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 2
Hepatic Cirrhosis (Hepatobiliary disorders) | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 1
Abscess Limb (Infections and infestations) | 2
Arthritis Infective (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Cholecystitis Infective (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 5
Haematoma Infection (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 4
Infectious Pleural Effusion (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lobar Pneumonia (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Lung Abscess (Infections and infestations) | 1
Muscle Abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Otitis Externa (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 22
Pyelonephritis Acute (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 6
Sepsis (Infections and infestations) | 6
Septic Shock (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 1
Soft Tissue Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 10
Vulval Abscess (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 2
Clavicle Fracture (Injury, poisoning and procedural complications) | 1
Compression Fracture (Injury, poisoning and procedural complications) | 1
Cranial Nerve Injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 5
Hip Fracture (Injury, poisoning and procedural complications) | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Patella Fracture (Injury, poisoning and procedural complications) | 2
Pelvic Fracture (Injury, poisoning and procedural complications) | 2
Pubis Fracture (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Arteriogram Coronary (Investigations) | 1
Blood Pressure Abnormal (Investigations) | 1
Ejection Fraction Decreased (Investigations) | 1
Electrocardiogram Abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 3
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Fistula (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1
Acute Lymphocytic Leukaemia Re (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Biliary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder Transitional Cell Carc (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pleural Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urethral Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid Artery Stenosis (Nervous system disorders) | 1
Cauda Equina Syndrome (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 7
Cognitive Disorder (Nervous system disorders) | 1
Complex Regional Pain Syndrome (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 2
Dizziness Postural (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hepatic Encephalopathy (Nervous system disorders) | 1
Loss Of Consciousness (Nervous system disorders) | 1
Neurodegenerative Disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 5
Transient Ischaemic Attack (Nervous system disorders) | 2
Viith Nerve Paralysis (Nervous system disorders) | 1
Confusional State (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Mental Disorder (Psychiatric disorders) | 1
Diabetic Nephropathy (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Prerenal Failure (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 6
Renal Failure Acute (Renal and urinary disorders) | 13
Renal Failure Chronic (Renal and urinary disorders) | 3
Urinary Retention (Renal and urinary disorders) | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2
Prostatomegaly (Reproductive system and breast disorders) | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Arteriovenous Fistula Operation (Surgical and medical procedures) | 1
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 1
Cataract Operation (Surgical and medical procedures) | 1
Colon Polypectomy (Surgical and medical procedures) | 1
Hip Arthroplasty (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 1
Limb Immobilisation (Surgical and medical procedures) | 1
Aortic Stenosis (Vascular disorders) | 6
Arteriovenous Fistula (Vascular disorders) | 2
Deep Vein Thrombosis (Vascular disorders) | 1
Femoral Arterial Stenosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 54
Hypertension (Vascular disorders) | 2
Hypertensive Crisis (Vascular disorders) | 6
Hypotension (Vascular disorders) | 1
Orthostatic Hypotension (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2
Peripheral Ischaemia (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 1
Vascular Stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE (N=963)
Anaemia (Blood and lymphatic system disorders) | 6
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2
Microcytic Anaemia (Blood and lymphatic system disorders) | 1
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Spontaneous Haematoma (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute Coronary Syndrome (Cardiac disorders) | 1
Angina Pectoris (Cardiac disorders) | 54
Atrial Fibrillation (Cardiac disorders) | 15
Atrial Flutter (Cardiac disorders) | 1
Atrial Thrombosis (Cardiac disorders) | 1
Atrioventricular Block Complete (Cardiac disorders) | 1
Atrioventricular Block First Degree (Cardiac disorders) | 3
Atrioventricular Block Second Degree (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 4
Bundle Branch Block Left (Cardiac disorders) | 2
Bundle Branch Block Right (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 7
Cardiac Failure Congestive (Cardiac disorders) | 1
Coronary Artery Dissection (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 8
Pericardial Effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Ventricular Tachycardia (Cardiac disorders) | 1
Phimosis (Congenital, familial and genetic disorders) | 1
Otorrhoea (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 8
Cataract (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Visual Impairment (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 4
Aphthous Stomatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Diverticulum (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Epigastric Discomfort (Gastrointestinal disorders) | 1
Gastric Disorder (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 8
Gastritis Erosive (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Inguinal Hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Peptic Ulcer (Gastrointestinal disorders) | 1
Tooth Loss (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chest Discomfort (General disorders) | 4
Chest Pain (General disorders) | 5
Fatigue (General disorders) | 3
Impaired Healing (General disorders) | 1
Nodule (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 4
Oedema (General disorders) | 3
Oedema Peripheral (General disorders) | 9
Pacemaker Generated Arrhythmia (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Spinal Pain (General disorders) | 1
Ulcer (General disorders) | 2
Biliary Colic (Hepatobiliary disorders) | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 1
Hepatic Steatosis (Hepatobiliary disorders) | 3
Liver Disorder (Hepatobiliary disorders) | 1
Asymptomatic Bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Enterobiasis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis Viral (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Lower Respiratory Tract Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Osteomyelitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Respiratory Tract Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tinea Cruris (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urethritis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 15
Vaginal Infection (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 6
Joint Injury (Injury, poisoning and procedural complications) | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 4
Wound (Injury, poisoning and procedural complications) | 1
Wound Complication (Injury, poisoning and procedural complications) | 1
Blood Calcium Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 2
Blood Glucose Abnormal (Investigations) | 1
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1
Cardiac Enzymes Increased (Investigations) | 1
Ejection Fraction Decreased (Investigations) | 2
Glycosylated Haemoglobin Increased (Investigations) | 1
Haemoglobin Decreased (Investigations) | 1
Prostatic Specific Antigen Increased (Investigations) | 1
Troponin I Increased (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 4
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 3
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Systemic Sclerosis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Balance Disorder (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 3
Cervicogenic Headache (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 9
Dizziness Postural (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 1
Petit Mal Epilepsy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Restless Legs Syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Transient Ischaemic Attack (Nervous system disorders) | 2
Tunnel Vision (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Listless (Psychiatric disorders) | 1
Sleep Disorder (Psychiatric disorders) | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 3
Nephrolithiasis (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 2
Renal Failure Acute (Renal and urinary disorders) | 6
Renal Failure Chronic (Renal and urinary disorders) | 3
Renal Impairment (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1
Vaginismus (Reproductive system and breast disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Rash Generalised (Skin and subcutaneous tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Cardiac Ablation (Surgical and medical procedures) | 1
Aortic Aneurysm (Vascular disorders) | 2
Arteriosclerosis (Vascular disorders) | 1
Femoral Arterial Stenosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 8
Haemorrhage (Vascular disorders) | 100
Hypertension (Vascular disorders) | 17
Hypertensive Crisis (Vascular disorders) | 4
Hypotension (Vascular disorders) | 5
Intermittent Claudication (Vascular disorders) | 1
Orthostatic Hypotension (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2
Vascular Dissection (Vascular disorders) | 1
Vascular Stenosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT03355742/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03355742/SAP_003.pdf